CLINICAL TRIAL: NCT05313802
Title: A Multiple Dose Study in Healthy Overweight and Obese Participants to Investigate the Safety, Tolerability, and Pharmacokinetics of LY3502970
Brief Title: A Study of LY3502970 in Healthy Overweight and Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18453; J2A-MC-GZGK (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-04-04; First posted 2022-04-06 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10-01

CONDITIONS: Healthy; Obese
Keywords: Pharmacokinetics; Safety and Tolerability; LY3502970
MeSH Terms: conditions — Obesity | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3502970 (Dose Level 1) (Experimental): LY3502970 administered orally.
  Interventions: Drug: LY3502970
- LY3502970 (Dose Level 2) (Experimental): LY3502970 administered orally.
  Interventions: Drug: LY3502970
- LY3502970 (Dose Level 3) (Experimental): LY3502970 administered orally.
  Interventions: Drug: LY3502970

INTERVENTIONS:
Drug: LY3502970 — Administered orally.

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3502970 in healthy overweight and obese participants. The blood tests will be conducted to measure how much LY3502970 is in the bloodstream and how the body handles and eliminates LY3502970 in these participants. The study will last up to 42 days excluding the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants with stable body weight for at least one month prior to randomization.
* Participants with body mass index (BMI) of greater than or equal to (≥) 27.0 kilograms per meter squared (kg/m²)
* Male participants who agree to use highly effective/effective methods of contraception and female participants not of childbearing potential

Exclusion Criteria:

* Have known allergies to LY3502970 or other glucagon-like peptide-1 Receptor Agonists (GLP-1 RA) analogs
* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological or neurological disorders
* Have any type of diabetes with hemoglobin A1c (HbA1c) ≥6.5 %

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Predose up to 42 days
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3502970 | Predose up to 29 days postdose
  PK: AUC of LY3502970
PK: Maximum Observed Concentration (Cmax) of LY3502970 | Predose up to 29 days postdose
  PK: Cmax of LY3502970
PK: Time to Maximum Observed Concentration (Tmax) of LY3502970 | Predose up to 29 days postdose
  PK: Tmax of LY3502970
Pharmacodynamics (PD): Change From Baseline in Body Weight | Predose through Day 28
  PD: Change From Baseline in Body Weight

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Qps-Mra, Llc, Miami, Florida
  - ICON Early Phase Services Lenexa Center, Lenexa, Kansas
  - ICON Early Phase Services, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No